CLINICAL TRIAL: NCT03236844
Title: A Multi-Center, Randomized, Open-Label, Single-Dose, Parallel Group Study to Investigate the Relative Bioavailability of Gantenerumab Produced With the G4 Process in Comparison to Gantenerumab Produced With the G3 Process Following Administration by Subcutaneous Injection in Healthy Volunteers
Brief Title: Relative Bioavailability of Gantenerumab Produced by G4 Process Versus G3 Process Following Subcutaneous (SC) Injection in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WP40052
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — gantenerumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gantenerumab G4 (Experimental): Participants will receive single dose of gantenerumab HCLF manufactured by G4 process on Day 1.
  Interventions: Drug: Gantenerumab
- Gantenerumab G3 (Experimental): Participants will receive single dose of gantenerumab HCLF manufactured by G3 process on Day 1.
  Interventions: Drug: Gantenerumab

INTERVENTIONS:
Drug: Gantenerumab — Gantenerumab HCLF manufactured by either G3 or G4 process will be administered on Day 1 (in the abdomen).
  Other Names: RO4909832

SUMMARY:
The purpose of this study is to assess the relative bioavailability of the high concentration liquid formulation (HCLF) of gantenerumab produced with the G4 process in comparison to the same HCLF of gantenerumab produced with the G3 process in healthy participants following single SC dose administration.

DETAILED DESCRIPTION:
This multi-center, randomized, open-label, single dose, parallel-group study will assess the relative bioavailability and the safety and tolerability of gantenerumab produced with the G4 process in comparison to gantenerumab produced with the G3 process. All participants will receive single SC dose of gantenerumab (manufactured by either the G3 or G4 process) on Day 1. The total duration of the study for each participant will be up to 21 weeks: Screening (up to 8 weeks); In-clinic period (Days -1 to 3); Out-patient period (Days 4 up to 68); and Safety Follow-up (up to 90 days after dosing).

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant
* Body mass index (BMI) between 18.0 and 30.0 kilograms per meter-square (kg/m^2), inclusive
* Body weight between 55 to 110 kg inclusive
* Female participants with either non-childbearing potential or with childbearing potential who commit to remain abstinent or use acceptable contraceptive methods during the treatment period and until at least 6 months after the follow-up visit
* Women of childbearing potential must have a negative serum pregnancy test result at screening and Day 1

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer, or cirrhosis
* History or suspicion of drugs of abuse addiction
* History or suspicion of alcohol addiction
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 17 weeks after the last dose of study drug
* Prior administration of gantenerumab
* Clinically significant abnormalities (as judged by the investigator) in laboratory test results (including complete blood count, chemistry panel, and urinalysis)
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the participant in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Gantenerumab | Predose (any time before injection), 1, 6, and 12 hours postdose (after injection) on Day 1; on Days 2, 3, 4, 5, 6, 7, 8, 12, 21, 29, 43, 64, and 85
Area Under the Plasma Concentration-Time Curve From Time Zero (Predose) to Extrapolated Infinite Time (AUC 0-inf) | Predose (any time before injection), 1, 6, and 12 hours postdose (after injection) on Day 1; on Days 2, 3, 4, 5, 6, 7, 8, 12, 21, 29, 43, 64, and 85

SECONDARY OUTCOMES:
Local Pain Assessments Using Visual Analog Scale (VAS) | After needle insertion, immediately postdose, 5 minutes (min), 10 min, 20 min, 1 hour, and 6 hours postdose on Day 1; on Days 2 and 3
Local Pain Assessments Using Verbal Rating Scale (VRS) | After needle insertion, immediately postdose, 5 min, 10 min, 20 min, 1 hour, and 6 hours postdose on Day 1; on Days 2 and 3
Skin Reactivity Assessment: Percentage of Participants by Severity of Injection Site Reactions | Immediately postdose, 10 min, 1 hour, and 6 hours postdose on Day 1; on Day 3
Skin Reactivity Assessment: Percentage of Participants by Size of Injection Site Reactions | Immediately postdose, 10 min, 1 hour, and 6 hours postdose on Day 1; on Day 3
Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | AEs: From Day 1 to Day 85; SAEs: From signing informed consent to end of study (maximum up to 5 months)
Percentage of Participants With Anti-Gantenerumab Antibodies | Predose (any time before injection) on Day 1 and on Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - PRA International Clinical Pharmacology Center (EDS US Clinic), Lenexa, Kansas
  - PRA, Marlton, New Jersey
  - PRA Health Sciences, Salt Lake City, Utah